CLINICAL TRIAL: NCT05809804
Title: Median Effective Dose of Esketamine Pretreatment to Prevent Sufentanil-induced Cough
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20230325
Record Dates: First submitted 2023-03-25; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Sufentanil; Esketamine
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Age range of 18 to 44 years olds (Experimental): The initial dose of esketamine was set as 0.06 mg / kg, and the injection time of esketamine was 5 s. One minute after injection of esketamine, sufentanil 0.4 μg / kg was injected within 5 s, and the number of coughs within 1 min after injection was recorded. According to the evaluation of sufentanil-induced cough, the dose of esketamine was adjusted. If the patient had no cough ( negative reaction ), the dose of esketamine in the next patient was reduced until the cough reaction occurred. If the patient had a cough reaction ( positive reaction ), the dose of esketamine in the next patient was increased until the cough disappeared. The dose ratio of adjacent esketamine was 1.1. Each group was selected from the previous patient with positive reaction until the 7 groups of positive and negative reactions appeared alternately, and the test was completed.
  Interventions: Drug: Esketamine
- Age range of 45 to 59 years olds (Experimental): The initial dose of esketamine was set as 0.06 mg / kg, and the injection time of esketamine was 5 s. One minute after injection of esketamine, sufentanil 0.4 μg / kg was injected within 5 s, and the number of coughs within 1 min after injection was recorded. According to the evaluation of sufentanil-induced cough, the dose of esketamine was adjusted. If the patient had no cough ( negative reaction ), the dose of esketamine in the next patient was reduced until the cough reaction occurred. If the patient had a cough reaction ( positive reaction ), the dose of esketamine in the next patient was increased until the cough disappeared. The dose ratio of adjacent esketamine was 1.1. Each group was selected from the previous patient with positive reaction until the 7 groups of positive and negative reactions appeared alternately, and the test was completed.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — The initial dose of esketamine was set as 0.06 mg / kg, and the injection time of esketamine was 5 s. One minute after injection of esketamine, sufentanil 0.4 μg / kg was injected within 5 s, and the number of coughs within 1 min after injection was recorded. According to the evaluation of sufentanil-induced cough, the dose of esketamine was adjusted. If the patient had no cough ( negative reaction ), the dose of esketamine in the next patient was reduced until the cough reaction occurred. If the patient had a cough reaction ( positive reaction ), the dose of esketamine in the next patient was increased until the cough disappeared. The dose ratio of adjacent esketamine was 1.1. Each group was selected from the previous patient with positive reaction until the 7 groups of positive and negative reactions appeared alternately, and the test was completed.

SUMMARY:
Sufentanil has the advantages of fast onset time, strong analgesic function and cardiovascular stability, and is widely used during general anesthesia induction. However, sufentanil can cause cough during induction of general anesthesia. Different studies have reported that the incidence of sufentanil-induced cough ( SIC ) during anesthesia is 16-42 %. This pathological condition may lead to damage to the central nervous system, increase the risk of reflux and aspiration, increase intracranial pressure and intraocular pressure, and endanger patients with cerebral aneurysms and ocular trauma. Therefore, at the moment of advocating comfortable anesthesia medical services, sufentanil-induced cough response is a problem that clinical anesthesiologists need to focus on and urgently solve. It has been reported that ketamine can reduce the incidence of cough caused by opioids. Esketamine is a pure dextro-enantiomer of ketamine and an NMDA antagonist with potent analgesic and bronchodilator effects. In this study, Dixon sequential method was used to study the median effective dose ( ED50 ) of intravenous esketamine pretreatment to prevent sufentanil-induced cough, and to explore the effect of age on ED50. To provide reference for clinical rational selection of esketamine dose.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II patients aged 18-59 years undergoing elective surgery under general anesthesia

Exclusion Criteria:

1. Preoperative intracranial pressure;
2. intra-abdominal pressure or intraocular pressure increased ;
3. have a history of cardiovascular and cerebrovascular diseases ;
4. have a history of asthma ;
5. have a history of chronic cough ;
6. have a history of smoking ;
7. there was a history of upper respiratory tract infection 2 weeks before operation;
8. Patients received opioid therapy 2 weeks before surgery.;
9. Patients who received angiotensin converting enzyme inhibitors, bronchodilators or steroids 2 weeks before surgery ;
10. abnormal liver and kidney function ; weight exceeded 20 % of the ideal weight ( male height - 100, female height - 105 ).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
The presence of cough | an average of 1 minutes
  Yes or No

SECONDARY OUTCOMES:
The levels of cough | an average of 1 minutes
  No cough: 0 times ; mild: 1-2 times ; moderate: 3-5 times ; severe: > 5 times